CLINICAL TRIAL: NCT05687448
Title: DIrect Oral Anticoagulant for Antithrombotic Management Of Aortic Bioprothesis Valve implaNted Patients for Valvular Heart Disease Study
Brief Title: DIrect Oral Anticoagulation and Bioprothesis Aortic Valve
Acronym: DIAMOND
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-516643-64-00
Record Dates: First submitted 2022-09-26; First posted 2023-01-18 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Disease
Keywords: Anticoagulant; Aortic valve; Apixaban; Aspirin; Stroke; Hemorrhage
MeSH Terms: conditions — Aortic Valve Disease; Stroke; Hemorrhage | interventions — apixaban; Tablets

STUDY DESIGN:
Intervention Model Description: This study is a national, multicentre, randomized, parallel-group, open label study in patients (aged ≥18 years) with aortic bioprosthesis at least 7 days after cardiac surgery.
  Experimental group:
  Patients treated with apixaban 5 mg twice daily (BID)
  Active Comparator group:
  Aspirin 75 to 100mg once a day
Masking Description: The Outcomes adjudication will be performed blinded of patients treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients treated with apixaban 5 mg twice daily (BID)
  Interventions: Drug: Apixaban 5 MG Oral Tablet
- Active Comparator group: (Active Comparator): Patients treated with Aspirin 75 to 100mg once a day
  Interventions: Drug: Aspirin 75 to 100mg once a day

INTERVENTIONS:
Drug: Apixaban 5 MG Oral Tablet — Patients treated with apixaban 5 mg twice daily (BID)
  Other Names: Experimental Group
  Arms: Experimental Group
Drug: Aspirin 75 to 100mg once a day — Patients treated with Aspirin 75 to 100mg once a day
  Other Names: Active Comparator
  Arms: Active Comparator group:

SUMMARY:
DIAMOND study is a national, multicentre, randomized, parallel-group, open label study in patients (aged ≥18 years) with aortic bioprosthesis (excluding TAVI) at least 7 days after cardiac surgery.

Experimental group:

Patients treated with apixaban 5 mg twice daily (BID)

Active Comparator group:

Aspirin 75 to 100mg once a day

The primary objective is to demonstrate that antithrombotic treatment with apixaban is superior to aspirin in patients with recent surgical bioprosthetic aortic valve replacement for the primary composite efficacy endpoint of death from any cause, myocardial infarction, stroke, systemic embolism, deep vein thrombosis, or pulmonary embolism and valve thrombosis after 105 days of follow-up.

DETAILED DESCRIPTION:
Early antithrombotic management of patients who have undergone aortic valve replacement using a bioprosthesis remains a source of medical concern. The optimal antithrombotic strategy early after surgery remains controversial due to lack of high-quality evidence. Some observational studies support the use of vitamin K antagonists (VKAs) compared to aspirin (ASA) to significantly reduce the risk of thromboembolism but suffer from major source of bias inherent to retrospective analyses of observational data. A small, randomized trial found that VKA for 3 months significantly increased major bleeding compared with ASA, without reducing the rate of deaths or thromboembolic events but this study was underpowered for ischemic events. There is therefore a lack of evidence demonstrating the superiority of anticoagulant treatment compared to aspirin early after bioprosthetic aortic valve surgery. Current ESC guidelines recommend that ASA or VKA should be considered for 3 months after surgical implantation of an aortic bioprosthesis. At the opposite, current AHA/ACC guidelines recommend that anticoagulation with VKA to achieve an INR of 2.5 is reasonable for at least 3 months and for as long as 6 months for patients at low risk of bleeding (IIa, level B). However, anticoagulation by VKAs is currently underused and guideline recommendations are not followed by most clinicians as VKAs have major drawbacks: narrow therapeutic window, variable dose-response in individuals, interaction with several foods and drugs.

Despite their superiority to reduce bleeding in patients with non-valvular atrial fibrillation compared to VKAs, direct oral anticoagulants (DOACs) including apixaban have not been well evaluated in the first 3 months after surgical bioprosthetic valve implantation. A small, randomized trial found that edoxaban was non-inferior to warfarin for preventing thromboembolism and the occurrence of major bleeding in the first 3 months after aortic or mitral surgical bioprosthetic valve implantation. DOAC(s) are effective in patients with atrial fibrillation and bioprosthetic valve implanted after 3 months.

Finally, there is an unmet clinical need for an alternative to ASA or VKAs, such as an anti-Xa DOAC like apixaban, as anticoagulation in patients in the first 3 months after surgical bioprosthetic valve implantation.

The purpose of this study is to compare the efficacy of apixaban and aspirin on ischemic endpoints during the first 3 months after aortic surgical bioprosthetic valve implantation excluding TAVI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Prior implantation of a surgical bioprosthesis in the aortic position at least 7 days and before hospital discharge (excluding TAVI)
3. Participants currently not requiring chronic anticoagulation for another reason (atrial fibrillation, pulmonary embolism or any other condition)
4. Patients affiliated to social security
5. Patient able to give free, informed and written consent

Exclusion Criteria:

1. Any cardiac surgery less than 7 days prior to enrollment or more than 1 month
2. Mechanical valve in any position or combined valve surgery (mitral or tricuspid).
3. Any major bleeding in the three months (90 days) prior to enrollment.
4. Active bleeding or high risk of bleeding after cardiac surgery (i.e. hemopericardium) or lesion or condition considered as a significant risk factor for major bleeding according to investigator
5. Atrial fibrillation requiring chronic anticoagulation
6. Need to be on dual antiplatelet therapy (aspirin >100 mg daily and a P2Y12 inhibitor, i.e. clopidogrel, ticagrelor, prasugrel) or requiring chronic anticoagulation whatever the treatment (oral or injection).
7. Known hypersensitivity or other contraindications to apixaban (hepatic disease associated with coagulopathy and clinically relevant bleeding risk).
8. Creatinine clearance <40 mL/min (Cockcroft) or patients requiring apixaban dose reduction.
9. Known hypersensitivity or other contraindications to aspirin (Hypersensitivity to aspirin or any of the excipients, history of asthma induced by the administration of salicylates, ongoing peptic ulcer, constitutional or acquired hemorrhagic disease including gastrointestinal bleeding, history of hemorrhagic stroke and thrombocytopenia, pregnancy after 24 weeks of gestation, risk of bleeding, severe renal failure, severe hepatic impairment, uncontrolled severe heart failure
10. Known hypersensitivity or other contraindications to heparin or low molecular weight heparin (history of heparin-induced thrombocytopenia, hypersensitivity to any of the excipients…)
11. Ischemic stroke within 1 month or intracranial hemorrhage
12. Active endocarditis at the time of screening for enrollment.
13. Women of childbearing potential without efficient contraception, pregnant or breastfeeding women.
14. Concomitant combined strong P-gp and CYP3A4 inducers or inhibitors.
15. History of non-compliance
16. Participation in another interventional study
17. Active cancer or life expectancy less than 1 year
18. Persons deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Clinical Events (MACE) | Up to 3.5 months
  The primary endpoint is a composite efficacy endpoint including death from any cause, myocardial infarction, stroke, systemic embolism, deep vein thrombosis, or pulmonary embolism and valve thrombosis.

SECONDARY OUTCOMES:
Bleeding | Up to 3.5 months
  ISTH major and non-major clinically relevant bleeding
Death | Up to 3.5 months
  Including cardiovascular and non cardiovascular death
Myocardial infarction | Up to 3.5 months
Stroke | Up to 3.5 months
Systemic embolism | Up to 3.5 months
Deep vein thrombosis or pulmonary embolism | Up to 3.5 months
Valve thrombosis | Up to 3.5 months
Bleeding | Up to 3.5 months
  According to ISTH major and non-major clinically relevant bleeding, BARC and TIMI 6, BARC and TIMI Classifications
Echographic parameter of aortic valve | Up to 3.5 months
  Variation of mean aortic gradient (mm/Hg)
Assessment of coagulation | Up to 3.5 months
  Measured by thrombin generation in a subgroup population (n=216)
To evaluate platelet activation (sP-selectin) in a subgroup population (n = 216) | Up to 3.5 months
To build a population PK/PD in the experimental group | Up to 3.5 months
  Measuring the apixaban concentration (anti-Xa activity expressed in ng/mL) (apixaban, n = 108)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Guillaume DILLINGER, Professor, Principal Investigator — Assistance Publique Hôpitaux Paris
Locations (1):
- Service de Cardiologie Hôpital Lariboisière, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No